CLINICAL TRIAL: NCT01078493
Title: Phase 1 Study of Intradermal Injection of Autologous Platelet Rich Plasma for Facial Wrinkles
Brief Title: Wrinkle Injection With Autologous Platelet Rich Plasma Study
Acronym: WIPES
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol revision necessary.
Sponsor: Novena Medical Center (Network)
Responsible Party: Dr Tan Kok Leong, Life Source Medical Centre @ Novena Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTC1000031
Record Dates: First submitted 2010-02-27; First posted 2010-03-02 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Wrinkles
Keywords: Platelet rich plasma; PRP; wrinkles; MyCells®; CREATE; Life Source Medical Centre; Dr Tan Kok leong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MyCells® (injection of platelet rich plasma) — PRP contains at least 1,000,000 platelets per mm3 or 2-6 times the native concentration of whole blood at a pH of 6.5 to 6.7
  Other Names: MyCells autologous platelet preparation system

SUMMARY:
Wrinkles result from imperfect repair of the dermal layer resulting in loss of collagen commonly due to ageing, smoking and sun exposure. Platelet rich plasma (PRP) contains a host of growth factors, which have been used in other clinical trials for various medical conditions such as tendonitis, and also in surgery such as the surgical repair of facial defects. Results from these clinical trials suggest that PRP helps in collagen formation and organisation to promote healing of tissues. This study attempts to document the clinical effects of intradermal injection of PRP on wrinkles.

DETAILED DESCRIPTION:
10 selected participants will have 10 ml of blood removed for platelet extraction with MyCells®. The resulting Platelet rich plasma will be injected intradermally into the facial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 21 years of age
* Dis-satisfied or anxious about facial wrinkles (total wrinkle length more than 1cm)

Exclusion Criteria:

* Pregnant women.
* Psychiatric patients.
* Known bleeding disorders such as platelet dysfunction syndrome, thrombocytopenia, hypofibrinogenemia
* Anticoagulants(eg.aspirin, warfarin)
* Had other wrinkle therapy for less than a month.(laser, peels, injections)
* Had facelift surgery for less than a year.
* Diseased states such as organ failure, severe anaemia, cancer, acute/chronic infections.
* Involved in personal litigation against an aesthetic service provider

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Total Wrinkle Length | 3 months
  All visible wrinkles are measured and the length is summed up to give the Total Wrinkle Length. Comparison of pre treatment and post treatment Total Wrinkle Length will be studied.

SECONDARY OUTCOMES:
Side effect / Adverse Event | 3 months
  Side Effects / Adverse Events to be monitored include allergic reaction, nerve injury and cavernous sinus thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kok Leong Tan, MBBS, Principal Investigator — Life Source Medical Centre @ Novena Medical Center
Locations (1):
- Life Source Medical Centre @ Novena Medical Center, Singapore, Singapore, Singapore